CLINICAL TRIAL: NCT05152082
Title: Establishment and Validation of a Predictive Model for the Risk of Colorectal Advanced Adenomas
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: 2021-SR-365
Record Dates: First submitted 2021-11-08; First posted 2021-12-09 (Actual); Last update posted 2021-12-30 (Actual); Status verified 2021-12

CONDITIONS: Colorectal Adenoma

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- patients with colorectal advanced adenomas
- patients without colorectal advanced adenomas

SUMMARY:
The study aimed to analyze the risk factors of colorectal advanced adenoma and constructe a model to predict the high-risk individuals of harbouring colorectal advanced adenomas, so as to better identify screening participants and provide an important theoretical basis for the prevention of colorectal cancer.

DETAILED DESCRIPTION:
A large cohort of eligible patients were included in the analysis, and classified into derivation and validation cohorts at a ratio of 7:3. Demographic and clinicopathological characteristics of participants were utilized to develop a prediction model for colorectal advanced polyps. In the derivation cohort, the LASSO regression method was applied to filter variables and multivariate logistic regression analysis was used to identify important predictors.A prediction model was established based on the results of multivariate logistic regression analysis. The predictive performance of the model was evaluated with respect to its discrimination, calibration and clinical usefulness.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged ≥18 and ≤75 years old. Patients with complete data on demography and clinicopathology.

Exclusion Criteria:

* Patients with a history of inflammatory bowel disease, enterophthisis, familial adenomatous polyposis, P-J syndrome and intestinal lymphoma.

Patients with a previous history of colorectal neoplasm. Patients with a history of severe systemic diseases. Lack of complete clinical data for analysis.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Confirmed eligible patients, 18 to 75 years of age, including cases with colorectal advanced adenomas and controls without colorectal advanced adenomas, are enrolled in this study.
Sampling Method: Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2021-06-01 (Actual); Primary Completion 2022-10-01 (Estimated); Study Completion 2022-12-01 (Estimated)

PRIMARY OUTCOMES:
Demographic characteristics of patients with colorectal adenomas checklist | 1 year
  Age (years), sex (man/woman), family history of colorectal cancer (in first-degree relatives, including parents and siblings), history of smoking (never, past, current), history of alcohol consumption (never, past, current), regular use of non-steroidal anti-inflammatory drugs
weight (kilograms) | 1 year
  Clinicopathological characteristics of patients with colorectal adenomas
height (meters) | 1 year
  Clinicopathological characteristics of patients with colorectal adenomas

SECONDARY OUTCOMES:
The important high-risk factors of colorectal advanced adenoma | 1 year
  The important high-risk factors with p value < 0.05

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital with Nanjing Medical University, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Betes M, Munoz-Navas MA, Duque JM, Angos R, Macias E, Subtil JC, Herraiz M, De La Riva S, Delgado-Rodriguez M, Martinez-Gonzalez MA. Use of colonoscopy as a primary screening test for colorectal cancer in average risk people. Am J Gastroenterol. 2003 Dec;98(12):2648-54. doi: 10.1111/j.1572-0241.2003.08771.x. PMID 14687811
- [Background] Wong MC, Lam TY, Tsoi KK, Hirai HW, Chan VC, Ching JY, Chan FK, Sung JJ. A validated tool to predict colorectal neoplasia and inform screening choice for asymptomatic subjects. Gut. 2014 Jul;63(7):1130-6. doi: 10.1136/gutjnl-2013-305639. Epub 2013 Sep 17. PMID 24045331